CLINICAL TRIAL: NCT02559791
Title: Route of Administration of Anti-IL5 Monoclonal Antibody in Prednisone-dependent Eosinophilic Asthma
Brief Title: Anti-Interleukin-5 (IL5) Monoclonal Antibody (MAb) in Prednisone-dependent Eosinophilic Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Teva Pharmaceuticals USA (Industry); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RES-38072
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2017-04

CONDITIONS: Severe Persistent Asthma; Eosinophilic Bronchitis
Keywords: Reslizumab; Eosinophils; Asthma; Airway inflammation; Prednisone
MeSH Terms: conditions — Asthma | interventions — reslizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study participants (Experimental): All study participants will receive 2 monthly doses of placebo followed by 4 monthly doses of IV reslizumab 3mg/kg
  Interventions: Biological: Reslizumab; Drug: Placebo

INTERVENTIONS:
Biological: Reslizumab — Reslizumab 3ml/kg once monthly for 4 months
  Other Names: Anti Il 5 monoclonal antibody
Drug: Placebo — Matching placebo once monthly for 2 months
  Other Names: 0.9% normal saline

SUMMARY:
The steroid sparing effect of anti interleukin (IL-5) monoclonal antibody has been proven, but the effectiveness of subcutaneous (SC) compared to intravenous (IV) administration of these drugs to suppress airway eosinophilia is still under debate. As part of a previous study, 100mg of mepolizumab were administered subcutaneously to a group of subjects with prednisone-dependent eosinophilic asthma. Despite this intervention, 50% of the subjects (15 patients participated in this study) had persistently elevated sputum eosinophil counts. The same 15 patients will be invited to participate in the current study, and if they provide their informed consent, will receive 2 monthly doses of placebo, followed by 4 monthly doses of IV reslizumab. The primary outcomes are blood and sputum eosinophils, and the secondary outcomes include sputum and blood Innate lymphoid cell-2 (ILC2) cells, cluster of differentiation 4 (CD4+) cells, cluster of differentiation-8 (CD8+) cells, cluster of differentiation-34 (CD34+), Eosinophil-Basophil cluster cells (Eo/B progenitor cells), forced expired volume in 1 second (FEV1), asthma control questionnaire (ACQ) and number of eosinophilic exacerbations. Measurements of the outcomes will be done before placebo, after placebo and after IV reslizumab. This study design will determine whether IV reslizumab is effective in suppressing airway eosinophilia in prednisone-dependent patients.

DETAILED DESCRIPTION:
Study design

Blinded placebo-controlled sequential clinical trial of 4 monthly doses of intravenously administered reslizumab.

The study will include two periods:

Period 1: After establishing the minimum dose of prednisone to observe sputum eosinophils ≥3% and blood eosinophils ≥300/µL, all subjects will receive 2 infusions (once monthly) of matching placebo.

Period 2: All subjects will then receive 4 infusions (once monthly) of reslizumab 3mg/kg.

Methods

15 patients (all of whom had sputum eosinophils ≥3% and blood eosinophils ≥300/µL) who were previously treated with S/C100 mg mepolizumab for at least 6 months, with the last dose at least 4 months before entering the study, will be invited to participate in the study.

Since discontinuing mepolizumab, these patients would have been re-established on their maintenance dose of daily prednisone + high doses of inhaled corticosteroids (ICS) and long acting beta agonist (LABA).

Baseline measurements of blood and sputum eosinophils, spirometry, symptoms (ACQ), and immune cells in blood and sputum (ILC2 cells, CD4 + cells, CD8+ cells, CD34+ Eo/B progenitor cells) will be enumerated by flow cytometry, and measures of local autoimmunity, using our established protocols at the start of Period 1 (baseline measurement).

They will then receive 2 infusions of placebo at monthly intervals, and measurements will be repeated at the end of Period 1 (post-placebo measurement).

The subjects will then receive by 4 infusions of 3 mg/kg reslizumab at monthly intervals. At the end of the 4 months, these measurements will be repeated (post-reslizumab measurement).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent Prior to the beginning of the study, patients must be willing and fully capable to provide written informed consent.
2. Prednisone-dependent eosinophilic asthma

   * Documented evidence of asthma: FEV1 reversibility of 12% and 200 ml after 200-400 micrograms of SABA. Or Methacholine challenge test <8mg/ml.
   * Documented history of persistent eosinophilia (sputum eosinophils ≥3% and/or blood eosinophils ≥300/µL) despite maintenance treatment with systemic glucocorticoids (5 to 35 mg per day of prednisone or its equivalent) before entering the study.
3. Previous treatment with 100 mg mepolizumab administered subcutaneously for at least 6 months, with the last dose at least 4 months before entering the study
4. Sputum eosinophils ≥3% and blood eosinophil ≥300/µL on visit 1 (screening visit).
5. Age between 18 and 75 years.
6. Male or eligible female subjects:

   To be eligible for entry into the study, females of childbearing potential (premenopausal women who are not permanently sterilized by means of hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) must commit to consistent and correct use of a highly effective method of birth control (true sexual abstinence, a vasectomized sexual partner, Implanon, female tubal occlusion, Intrauterine device (IUD), Depo provera injections, oral contraceptive pills or Nuvaring) for the duration of the trial and for 3 months after the last study drug administration. A serum pregnancy test is required of all females at the initial Baseline Visit (Visit 1). In addition, a urine pregnancy test will be performed for all females prior to enrollment, during each scheduled study visit prior to the injection of investigational product, and during the Follow-up Visit.
7. Male subjects who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of study drug and for 3 months after the last dose of study drug.

Exclusion Criteria:

1. Currently receiving another monoclonal antibody
2. Currently receiving other investigational drug or immunosuppressive medication
3. Known hypersensitivity to Reslizumab product or any of its excipients.
4. Intolerance, hypersensitivity, insensitivity or neutralizing antibody to mepolizumab.
5. Malignancy within the last 2 years
6. Any co-morbidity that the investigator believes is a contraindication. This includes but is not limited to any respiratory (eg. COPD, pulmonary fibrosis, EGPA, ABPA), cardiovascular, gastrointestinal, hematological, neurological, immunological, musculoskeletal, renal, infectious, neoplastic or inflammatory condition that may place the safety of the subject at risk during the duration of the study, influence the results of the study or their interpretation, or prevent the patient from completing the entire duration of the study.
7. Current pregnancy or lactation
8. Current smoker or ex-smoker with a smoking history greater than 20 pack years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophil percentage | Measured before the placebo phase (week 2), after 2 infusions of placebo (week 10), and after 4 infusions (week 26) of reslizumab 3mg/kg
  Change in sputum eosinophil %
Blood eosinophil absolute number | Measured before the placebo phase (week 2), after 2 infusions of placebo (week 10), and after 4 infusions/4 months (week 26) of reslizumab 3mg/kg
  Change in blood eosinophil absolute number

SECONDARY OUTCOMES:
Sputum and blood blood Innate lymphoid cell-2 (ILC2) cells, cluster of differentiation 4 (CD4+) cells, cluster of differentiation-8 (CD8+) cells, cluster of differentiation-34 (CD34+), Eosinophil-Basophil cluster cells (Eo/B progenitor cells), | Measured before the placebo phase (week 2), after 2 infusions of placebo (week 10), and after 4 infusions (week 26)of reslizumab 3mg/kg
  Change in absolute number of both sputum and blood blood Innate lymphoid cell-2 (ILC2) cells. Change in absolute number of different T-lymphocyte populations in cluster of differentiation 4 (CD4+) cells, cluster of differentiation-8 (CD8+) cells, cluster of differentiation-34 (CD34+) and Eosinophil-Basophil cluster cells (Eo/B progenitor cells),
Forced Expiratory Volume in 1 second (FEV1) | Measured before the placebo phase (week 2), after 2 infusions of placebo (week 10), and after 4 infusions (week 26) of reslizumab 3mg/kg
  Change in Forced Expiratory Volume in 1 second (FEV1)
Asthma Control Questionnaire (ACQ) | Measured before the placebo phase (week 2), after 2 infusions of placebo (week 10), and after 4 infusions (week 26) of reslizumab 3mg/kg
  Change in ACQ
Number of eosinophilic exacerbations | During the placebo phase (2 months/weeks 2-10) and during the Reslizumab phase (weeks 10-26) 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] D'silva L, Cook RJ, Allen CJ, Hargreave FE, Parameswaran K. Changing pattern of sputum cell counts during successive exacerbations of airway disease. Respir Med. 2007 Oct;101(10):2217-20. doi: 10.1016/j.rmed.2007.05.010. Epub 2007 Jul 2. PMID 17606366
- [Background] Nair P, Dasgupta A, Brightling CE, Chung KF. How to diagnose and phenotype asthma. Clin Chest Med. 2012 Sep;33(3):445-57. doi: 10.1016/j.ccm.2012.05.003. Epub 2012 Jul 7. PMID 22929094
- [Background] Bousquet J, Mantzouranis E, Cruz AA, Ait-Khaled N, Baena-Cagnani CE, Bleecker ER, Brightling CE, Burney P, Bush A, Busse WW, Casale TB, Chan-Yeung M, Chen R, Chowdhury B, Chung KF, Dahl R, Drazen JM, Fabbri LM, Holgate ST, Kauffmann F, Haahtela T, Khaltaev N, Kiley JP, Masjedi MR, Mohammad Y, O'Byrne P, Partridge MR, Rabe KF, Togias A, van Weel C, Wenzel S, Zhong N, Zuberbier T. Uniform definition of asthma severity, control, and exacerbations: document presented for the World Health Organization Consultation on Severe Asthma. J Allergy Clin Immunol. 2010 Nov;126(5):926-38. doi: 10.1016/j.jaci.2010.07.019. PMID 20926125
- [Background] Green RH, Brightling CE, McKenna S, Hargadon B, Parker D, Bradding P, Wardlaw AJ, Pavord ID. Asthma exacerbations and sputum eosinophil counts: a randomised controlled trial. Lancet. 2002 Nov 30;360(9347):1715-21. doi: 10.1016/S0140-6736(02)11679-5. PMID 12480423
- [Background] Jayaram L, Pizzichini MM, Cook RJ, Boulet LP, Lemiere C, Pizzichini E, Cartier A, Hussack P, Goldsmith CH, Laviolette M, Parameswaran K, Hargreave FE. Determining asthma treatment by monitoring sputum cell counts: effect on exacerbations. Eur Respir J. 2006 Mar;27(3):483-94. doi: 10.1183/09031936.06.00137704. PMID 16507847
- [Background] Nissim Ben Efraim AH, Levi-Schaffer F. Tissue remodeling and angiogenesis in asthma: the role of the eosinophil. Ther Adv Respir Dis. 2008 Jun;2(3):163-71. doi: 10.1177/1753465808092281. PMID 19124368
- [Background] Zhang J, Kuvelkar R, Murgolo NJ, Taremi SS, Chou CC, Wang P, Billah MM, Egan RW. Mapping and characterization of the epitope(s) of Sch 55700, a humanized mAb, that inhibits human IL-5. Int Immunol. 1999 Dec;11(12):1935-44. doi: 10.1093/intimm/11.12.1935. PMID 10590259
- [Background] Haldar P, Brightling CE, Hargadon B, Gupta S, Monteiro W, Sousa A, Marshall RP, Bradding P, Green RH, Wardlaw AJ, Pavord ID. Mepolizumab and exacerbations of refractory eosinophilic asthma. N Engl J Med. 2009 Mar 5;360(10):973-84. doi: 10.1056/NEJMoa0808991. PMID 19264686
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Ortega HG, Liu MC, Pavord ID, Brusselle GG, FitzGerald JM, Chetta A, Humbert M, Katz LE, Keene ON, Yancey SW, Chanez P; MENSA Investigators. Mepolizumab treatment in patients with severe eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1198-207. doi: 10.1056/NEJMoa1403290. Epub 2014 Sep 8. PMID 25199059
- [Background] Castro M, Mathur S, Hargreave F, Boulet LP, Xie F, Young J, Wilkins HJ, Henkel T, Nair P; Res-5-0010 Study Group. Reslizumab for poorly controlled, eosinophilic asthma: a randomized, placebo-controlled study. Am J Respir Crit Care Med. 2011 Nov 15;184(10):1125-32. doi: 10.1164/rccm.201103-0396OC. Epub 2011 Aug 18. PMID 21852542
- [Background] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060
- [Background] Nair P, Pizzichini MM, Kjarsgaard M, Inman MD, Efthimiadis A, Pizzichini E, Hargreave FE, O'Byrne PM. Mepolizumab for prednisone-dependent asthma with sputum eosinophilia. N Engl J Med. 2009 Mar 5;360(10):985-93. doi: 10.1056/NEJMoa0805435. PMID 19264687
- [Background] Nair P. Anti-interleukin-5 monoclonal antibody to treat severe eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1249-51. doi: 10.1056/NEJMe1408614. Epub 2014 Sep 8. No abstract available. PMID 25197762
- [Background] McKenzie AN. Type-2 innate lymphoid cells in asthma and allergy. Ann Am Thorac Soc. 2014 Dec;11 Suppl 5(Suppl 5):S263-70. doi: 10.1513/AnnalsATS.201403-097AW. PMID 25525730
- [Background] Hogan SP, Rosenberg HF, Moqbel R, Phipps S, Foster PS, Lacy P, Kay AB, Rothenberg ME. Eosinophils: biological properties and role in health and disease. Clin Exp Allergy. 2008 May;38(5):709-50. doi: 10.1111/j.1365-2222.2008.02958.x. Epub 2008 Apr 1. PMID 18384431
- [Background] Smith SG, Chen R, Kjarsgaard M, Huang C, Oliveria JP, O'Byrne PM, Gauvreau GM, Boulet LP, Lemiere C, Martin J, Nair P, Sehmi R. Increased numbers of activated group 2 innate lymphoid cells in the airways of patients with severe asthma and persistent airway eosinophilia. J Allergy Clin Immunol. 2016 Jan;137(1):75-86.e8. doi: 10.1016/j.jaci.2015.05.037. Epub 2015 Jul 17. PMID 26194544
- [Background] Kabata H, Moro K, Fukunaga K, Suzuki Y, Miyata J, Masaki K, Betsuyaku T, Koyasu S, Asano K. Thymic stromal lymphopoietin induces corticosteroid resistance in natural helper cells during airway inflammation. Nat Commun. 2013;4:2675. doi: 10.1038/ncomms3675. PMID 24157859
- [Derived] Mukherjee M, Aleman Paramo F, Kjarsgaard M, Salter B, Nair G, LaVigne N, Radford K, Sehmi R, Nair P. Weight-adjusted Intravenous Reslizumab in Severe Asthma with Inadequate Response to Fixed-Dose Subcutaneous Mepolizumab. Am J Respir Crit Care Med. 2018 Jan 1;197(1):38-46. doi: 10.1164/rccm.201707-1323OC. PMID 28915080
- See also: Global Initiative for Asthma. GINA report, global strategy for asthma management and prevention. Report 2015. — http://www.ginasthma.org.